CLINICAL TRIAL: NCT04321707
Title: Complete Local Response to Neoadjuvant Chemotherapy in Patients With Muscle Invasive Bladder Cancer Evaluated by 15O-H2O PET/MR
Acronym: MAINTAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jørgen Bjerggaard Jensen (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Consultant, MD, DMSc, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MAINTAIN
Record Dates: First submitted 2020-03-11; First posted 2020-03-25 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
Keywords: Tumor blood flow; magnetic resonans imaging; 15O water PET
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, explorative, single arm, non-randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 15O-H2O PET/MR (Experimental): All included patients will have two 15O-H2O PET/MR scan performed.
  Interventions: Radiation: 15O-H2O PET/MR

INTERVENTIONS:
Radiation: 15O-H2O PET/MR — All included patients will have a 15O-H2O PET/MR scan performed at baseline and a scan performed after NAC, prior to cystectomy.

SUMMARY:
Treatment of localized muscle invasive bladder cancer (MIBC) is radical cystectomy. Neoadjuvant chemotherapy (NAC) improves survival.

Approximately 50-60% of all MIBC patients undergoing NAC before cystectomy are histopathological without remnant tumor in the cystectomy specimen (T0). However, there is currently no optimal method to evaluate whether the patient is true T0 or has remnant tumor in need for consolidating radical treatment. The study aim is to investigate if 15O-H2O PET/MR can predict complete local response to neoadjuvant chemotherapy in patients with MIBC and thereby identify potential candidates for organ preservation.

DETAILED DESCRIPTION:
For patients with MIBC treated with NAC and radical cystectomy there is currently no good way of evaluating whether the patient is true T0 or has remnant tumor in need for consolidating radical treatment. Methods for better selection of patients that potentially can avoid cystectomy is therefore needed.

15O-labeled water (H2O) is the gold standard for PET quantification of regional tissue perfusion. 15O-H2O has been validated as a freely diffusible tracer for measuring perfusion in the myocardium and cerebral blood flow and 15O-H2O PET is the golden standard for noninvasive imaging to quantify tumor blood flow (TBF).

Method: Patients scheduled for NAC followed by radical cystectomy due to histologically documented MIBC stage cT2-4a in the urinary bladder will be included. A 15O-H2O PET/MR scan will be performed at time of inclusion (baseline) and again after NAC prior to cystectomy.

Hypothesis: We hypothesize that changes in tumor architecture and perfusion estimated with 15O-H2O PET/MR measurements and clinical evaluation during NAC can identify patients with complete local response to chemotherapy and therefore select patients to avoid radical cystectomy.

Perspectives: This study will be the first to use 15O-H2O as tracer in bladder cancer. If proven efficient, evaluation of patients undergoing NAC with 15O-H2O PET/MR could potentially safely select patients for a true bladder sparring approach and potentially give some patients the choice of chemotherapy monotherapy, or in combination with other systemic oncological treatments like immunotherapy. If successful, this should be followed by randomized studies to document the clinical benefit and potentially reduce cost and increase quality of life by safely selecting patients for bladder sparring treatment of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MIBC stage cT2-4a.
* Preoperative PET/CT of thorax, abdomen, and pelvis with no suspicion of organ metastases or lymph node metastasis outside the surgical field.
* ≥18 years of age at the time of signing the Informed Consent Form. Renal function of eGFR > 60 ml/min/1,73 m2.
* Physically fit for NAC.
* Clinical decision with patient accept of NAC before cystectomy.
* Mentally healthy. Signed Informed Consent Form.

Exclusion Criteria:

- Unfit for MRI:

* Claustrophobia.
* Problems with seating arrangements (e.g. pain or involuntary movement).
* Maximal shoulder width larger than 55 cm.
* Circumference larger than 160 cm.
* Weight above 250 kg.
* Metallic implants or other metallic foreign bodies.
* Pacemaker, ICD, or pace electrodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in tumor blood flow | Comparison of scan made 1 week before NAC compared to scan 2 weeks after NAC
  Change in Tumor Blood Flow (TBF) measured on 15O-H2O PET/MR as a marker of response to NAC correlated with histopathological findings in the cystectomy specimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Aarhus University Hopsital, Aarhus, Denmark